CLINICAL TRIAL: NCT04810741
Title: Retrospective Study of Clinical Practice and Management of Imported Schistosomiasis in France
Acronym: RETROBIZH
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201071
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2021-03

CONDITIONS: Schistosomiasis
Keywords: schistosomiasis, retrospective
MeSH Terms: conditions — Schistosomiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Schistosomiasis is a major public health issue. Clinical guidelines for the management of imported schistosomiasis are heterogeneous. The objective of this study is to describe the clinical management of schistosomiasis imported cases in France, regarding diagnosis, treatment and follow-up.

DETAILED DESCRIPTION:
Schistosomiasis is a major public health issue. Clinical guidelines for the management of imported schistosomiasis are heterogeneous. The objective of this study is to describe the clinical management of schistosomiasis imported cases in France, regarding diagnosis, treatment and follow-up. It is a multicentric, retrospective, descriptive study. Inclusion criteria are an age ≥ 18, a positive western blot and / or a positive microscopy exam. Data concerning clinical presentation, biological samples, imaging, treatment and follow-up will be assessed. A descriptive analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18, positive schistosomiasis immunoblot and / or positive microscopy examination for schistosomiasis eggs

Exclusion Criteria:

* - patients under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years-old with a diagnosis of schistosomiasis in France
Sampling Method: Non-Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Describe the management of patients with chronic schistosomiasis in France, in terms of diagnosis, assessment, management and follow-up. | 12 months
  Draft of new clarified recommendations on the overall management of this pathology

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Jareguiberry, Professor, Principal Investigator — APHP
Locations (1):
- hospital BICETRE, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No
No sharing